CLINICAL TRIAL: NCT01196260
Title: Clinical Trial on Combination Chemotherapy Treatments in Patients With Colorectal Cancer Stage II and III Among Chinese Population
Brief Title: Combination Chemotherapy Treatments in Patients With Colorectal Cancer Stage II and III
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Cancer Biology (Network)
Collaborators: Tianjin Union Medical Center (Other); Beihua University (Other); Chengdu Medical College (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Dake Chu, Dr., State Key Laboratory of Cancer Biology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dake Chu-200401; StateKeyLab (Registry Identifier: StateKeyLab)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
Keywords: efficiency; capecitabine; oxaliplatin; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-fluorouracil plus oxaliplatin (Experimental): patients will be randomized assigned to receive 5-fluorouracil plus oxaliplatin
  Interventions: Drug: Capecitabine and Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine and Oxaliplatin — Capecitabine and Oxaliplatin will be under the NSCLC guideline
  Other Names: 1220099; CDK

SUMMARY:
This study will examine a new combination of drugs: Capecitabine and Oxaliplatin for the treatment of Stage II and III colorectal cancer. Capecitabine and Oxaliplatin are approved by the Food and Drug Administration (FDA) for use in colorectal cancer. The combination of drugs is experimental (not approved by the FDA as standard treatment), but is a widely used treatment option and preliminary studies have shown that treatment with the combination has a positive effect on metastatic colorectal cancer.

DETAILED DESCRIPTION:
This study will examine a new combination of drugs: Capecitabine and Oxaliplatinfor for the treatment of Stage II and III colorectal cancer. Capecitabine and Oxaliplatin are approved by the Food and Drug Administration (FDA) for use in colorectal cancer. The combination of drugs is experimental (not approved by the FDA as standard treatment), but is a widely used treatment option and preliminary studies have shown that treatment with the combination has a positive effect on metastatic colorectal cancer. In the present trial, we will study the combination of these two drugs in patients with colorectal cancer among Chinese population

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically proven TNM stage II or III adenocarcinoma of colon or rectum.
* Patient must received curative surgical with cancer free margin.
* Patients must have a performance status of 0,1, or 2.
* Patients must have an absolute neutrophil count of greater than or equal to 1500/ml, platelet count greater than or equal to 100,000/ml, and total serum bilirubin equal or less than the institution's upper limit or normal range.
* Patients must have fully recovered from any effects of surgery.
* Patients must provide a signed consent to participate in the study.

Age:

•18 and over

Performance status:

•WHO 0-2

Life expectancy:

•Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 1.5 times ULN

Renal:

•Creatinine clearance greater than 30 mL/min

Cardiovascular:

More than 12 months since prior and no active clinically significant cardiovascular disease, including any of the following:

* Cerebrovascular accident
* Myocardial infarction
* Unstable angina
* New York Heart Association class II-IV congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active peptic ulcer or gastrointestinal bleeding within the past year
* No inflammatory bowel disease
* No other malignancy within the past 10 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

Exclusion Criteria:

* Patients with a proven history of peptic ulcer disease or gastroesophageal reflux.
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other non-steroidal anti-inflammatory drugs.
* Patients who have received prior chemotherapy for colorectal cancer except for patients relapsing more than 6 months after completion of adjuvant chemotherapy.
* History of other malignancy, except for cancers that have been treated with a curative intent and patient is without evidence of active disease.
* Unresolved bacterial infection requiring treatment with antibiotics.
* Pregnant or lactating women may not participate in the study. Women/men of reproductive age group may not participate unless they have agreed to use an effective method of contraception.
* Patients who have allergy to any of the study drugs.
* Patients known to have HIV-1 virus infection because of the undetermined effect of this chemotherapy regimen in patients with HIV-1 and the potential for serious interaction with anti-HIV medications.
* Gilbert's disease.
* Lack of physical integrity of the upper gastrointestinal tract. Inability to swallow tablets or those who have malabsorption syndrome.
* Other serious concurrent infection
* Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2004-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To determine the objective response rate of patients with metastatic colorectal cancer received the combination of drugs | 7 years
To determine the relapse of patients with metastatic colorectal cancer received the combination of drugs | 7 years
To determine prognosis of patients with metastatic colorectal cancer received the combination of drugs | 7 years

SECONDARY OUTCOMES:
To evaluate the time to progression of metastatic colorectal cancer after treatment | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Dake Chu, M.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- State Key Laboratory of Cancer Biology, Xi'an, Shaanxi, China

REFERENCES:
- See also: Related Info — http://www.fmmu.edu.cn